CLINICAL TRIAL: NCT00801996
Title: Epidemiologic, Clinical and Genetic Profile of Prostate Cancer in Arab Countries
Acronym: ProstateCA
Status: Withdrawn | Type: Observational
Why Stopped: Closed by Investigator
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0806009874
Record Dates: First submitted 2008-11-14; First posted 2008-12-04 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; genetics
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and tissue will be collected from individuals with prostate cancer. Only blood will be collected from normal controls.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. Prostate Cancer: Inclusion Criteria:
  * All study subjects should be able to provide informed consent
  * Males ages 40 years or older
  * Individuals from the Qatari Peninsula whose ancestors up to three generations back were natives of Qatar.
  * Individuals undergoing Trans Rectal Ultrasound (TRUS) biopsy as dictated by their standard clinical care
  * Ultrasound OR digital rectal examination consistent with prostate disease OR A level of PSA (Prostatic Specific Antigen) greater than 3.0
  Exclusion Criteria:
  • Patient refuses consent
- 2. Normal Healthy Controls: Inclusion Criteria:
  * All study subjects should be able to provide informed consent
  * Males or females ages 40 years or older (see section A8 for the rationale for the inclusion of females)
  * Individuals of Arab descent from Qatari peninsula without any personal or family history of prostate cancer
  Exclusion Criteria:
  * Individuals with family history of prostate cancer
  * Individuals not deemed in good overall health by the investigator will not be accepted into the study

SUMMARY:
This protocol is designed to collect a small amount of blood and tissue from individuals with prostate cancer for extraction of DNA (genetic material) for the study of the genetic basis of prostate cancer. The study population will include individuals with known prostate cancer and controls without prostate cancer. The study will be conducted in Doha, Qatar at the Hamad Medical Corporation and Weill Cornell Medical College (Qatar). Individuals in the study population will be of Arab descent from Qatar. In this protocol, researchers will survey epidemiologic factors and medical records of patients with prostate cancer in order to study the clinical characteristics of these individuals. The researchers will collect blood and tissue samples to evaluate the genetic characteristics of individuals with prostate cancer. The researchers will also collect blood samples of individuals without prostate cancer to serve as a control. The goal will be to identify genes that are associated with prostate cancer and gene profiles that are associated with differing prognoses in individuals who have prostate cancer.

DETAILED DESCRIPTION:
The study population will include individuals with known prostate cancer and controls without prostate cancer. Individuals in the study population will be of Arab descent from Qatar. In this protocol, researchers will survey epidemiologic factors and medical records of patients with prostate cancer in order to study the clinical characteristics of these individuals. The researchers will collect blood and tissue samples to evaluate the genetic characteristics of individuals with prostate cancer. The researchers will also collect blood samples of individuals without prostate cancer to serve as a control. The goal will be to identify genes that are associated with prostate cancer and gene profiles that are associated with differing prognoses in individuals who have prostate cancer.

ELIGIBILITY:
Inclusion/Exclusion Criteria for Normal Cohort

Inclusion Criteria:

* All study subjects should be able to provide informed consent
* Males or females ages 40 years or older (see section A8 for the rationale for the inclusion of females)
* Individuals of Arab descent from Qatari peninsula without any personal or family history of prostate cancer

Exclusion Criteria:

* Individuals with family history of prostate cancer
* Individuals not deemed in good overall health by the investigator will not be accepted into the study

Inclusion/Exclusion Criteria for Prostate Cohort

Inclusion Criteria:

* All study subjects should be able to provide informed consent
* Males ages 40 years or older
* Individuals from the Qatari Peninsula whose ancestors up to three generations back were natives of Qatar.
* Individuals undergoing Trans Rectal Ultrasound (TRUS) biopsy as dictated by their standard clinical care
* Ultrasound OR digital rectal examination consistent with prostate disease OR A level of PSA (Prostatic Specific Antigen) greater than 3.0

Exclusion Criteria:

• Patient refuses consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Individuals of Arab descent from Qatari peninsula
  * Individuals from the Qatari Peninsula whose ancestors up to three generations back were natives of Qatar
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Identification of single nucleotide polymorphisms (SNPs) in genes associated with prostate cancer in the Qatari population. | 3 years

SECONDARY OUTCOMES:
Use of gene expression profiles to develop molecular signatures of prostate cancer that are associated with clinical/pathological phenotypes (e.g., tumor grade, histology, disease stage, responsiveness to therapy) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Crystal, MD, Study Director — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College - Qatar, Doha, Qatar, Qatar

IPD SHARING:
Plan to Share IPD: Undecided